CLINICAL TRIAL: NCT06327516
Title: Lysophosphatidylglycerol in Asthma Pathogenesis
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020023
Record Dates: First submitted 2024-03-17; First posted 2024-03-25 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Asthma
Keywords: asthma; lysophosphatidylglycerol; Treg
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to investigate the relationship between the small molecule metabolite lysophosphatidylglycerol and asthma clinical features and explore its involvement in asthma pathogenesis.

DETAILED DESCRIPTION:
This study screened LPG as a asthma marker by performing metabolomics of the included asthma patients and normal controls, explored the relationship between LPG and clinical features of asthma (including acute exacerbation, asthma control state, asthma treatment steps，lung function, and inflammatory signals including eosinophils, FeNO and total IgE), and further performed in vitro tests to investigate the specific mechanism of LPG's involvement in asthma inflammation through its influence on Treg function.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of asthma.

Exclusion Criteria:

1. Combined with chronic obstructive pulmonary disease, bronchiectasis, pneumonia, obstructive sleep apnea hypopnea syndrome, malignant tumor
2. Combined with acute and chronic respiratory failure
3. Combined with severe cardiovascular disease
4. Pregnant woman.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with asthma who visited or were hospitalized in the Department of Respiratory and Critical Care Medicine of Peking University Third Hospital, who met the asthma diagnostic criteria proposed in the Bronchial Asthma Prevention and Treatment Guidelines and healthy controls without history or symptoms of chronic respiratory disease, allergic status or other conditions that could affect the outcome.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
lipidomics | when enrolled
  collect blood for lipidomic analysis and in vitro assays on Day1

CONTACTS AND LOCATIONS:
Overall Officials: Chun Chang, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking university third hospital, Beijing, None Selected, China

IPD SHARING:
Plan to Share IPD: Undecided